CLINICAL TRIAL: NCT00901238
Title: Intra-arterial Chemotherapy(Chemosurgery) for Retinoblastoma
Acronym: Chemosurgery
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: David Abramson,MD, Weill Cornell Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RTB1
Record Dates: First submitted 2009-05-12; First posted 2009-05-13 (Estimated); Last update posted 2009-12-17 (Estimated); Status verified 2009-12

CONDITIONS: Retinoblastoma
Keywords: retinoblastoma; intra-arterial chemotherapy; chemosurgery; melphalan; topotecan
MeSH Terms: conditions — Retinoblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Intra-arterial Chemotherapy — selective catheterization of the ophthalmic artery and injection of melphalan and topotecan
  Other Names: chemosurgery

SUMMARY:
Conventional treatments of retinoblastoma involves laser photocoagulation, cryotherapy (freezing of the tumor), plaque radiotherapy,external beam radiotherapy, and intravenous chemotherapy. Enucleation (removing of the eye)is the last option when the tumor cannot be controlled otherwise. However,many children with retinoblastoma present with advanced intraocular disease for which enucleation is the only option. Intra-arterial chemotherapy (Chemosurgery)delivers anti-tumor drug directly into the ophthalmic artery (the artery feeding the eye) in order to increase the dose of drug reaching the tumor while minimizing toxicity to the rest of the body.

DETAILED DESCRIPTION:
Present treatments for intraocular retinoblastoma cure 99% of children but have significant toxicity. Enucleation of the eye is effective but blinds the eye and leaves a lifelong cosmetic deformity. Radiation is associated with the subsequent development of fatal cancers. Systemic (intravenous)chemotherapy is used worldwide but experience with it has shown that the majority of eyes initially treated with chemotherapy still require additional treatments, such as radiation, laser, cryotherapy or even enucleation. In addition blood transfusions, secondary infections, insertion of ports and permanent hearing loss are now well reported. Three years ago we developed this technique of Chemosurgery for significantly increasing the dose of drug to the cancer while decreasing the dose of drug administered to children. This approach has decreased the need for enucleation in advanced eyes scheduled for enucleation with minimal systemic toxicity. We now offer treatment of both eyes simultaneously (in bilateral cases) and to eyes with less advanced disease and normal vision as an alternative to toxic systemic chemotherapy. In cases of very advanced ocular disease we will be using multiple drugs infused at the same session to increase tumor kill.

Chemosurgery interventions are performed under general anesthesia. The femoral artery (artery at the groin) is punctured and a catheter (a small plastic tube)is advanced into the opthalmic artery (the artery of the eye)using fluoroscopic (X-ray) guidance. The drugs are injected directly into the opthalmic artery over a period of 30-45 min.The catheter is then removed, manual compression exerted to the femoral artery, the child is awaken and goes to recovery for 6 hours. The procedure is repeated every 3-4 weeks for a total of 2 to 6 sessions according to tumor response. Since April 2006, our center has treated by chemosurgery 60 eyes in 52 patients with advanced intra-ocular retinoblastoma for which enucleation was considered.

ELIGIBILITY:
Inclusion Criteria:

* advanced retinoblastoma in one or both eyes
* recurrent retinoblastoma after failure of conventional methods

Exclusion Criteria:

* retinoblastoma judged curable by conventional methods
* patient judged unable to undergo the procedure

Min Age: 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2006-05; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
tumor control | 6 month

SECONDARY OUTCOMES:
tumor control with vision | 6 month

CONTACTS AND LOCATIONS:
Overall Officials: David H Abramson, MD, Principal Investigator — Weill Cornell Medical College and Memorial Sloan-Kettering Cancer Center
Locations (2):
- United States (2):
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Weill Medical College of Cornell University, New York, New York

REFERENCES:
- [Background] Brodie SE, Pierre Gobin Y, Dunkel IJ, Kim JW, Abramson DH. Persistence of retinal function after selective ophthalmic artery chemotherapy infusion for retinoblastoma. Doc Ophthalmol. 2009 Aug;119(1):13-22. doi: 10.1007/s10633-008-9164-3. Epub 2009 Jan 25. PMID 19169884
- [Result] Abramson DH, Dunkel IJ, Brodie SE, Kim JW, Gobin YP. A phase I/II study of direct intraarterial (ophthalmic artery) chemotherapy with melphalan for intraocular retinoblastoma initial results. Ophthalmology. 2008 Aug;115(8):1398-404, 1404.e1. doi: 10.1016/j.ophtha.2007.12.014. Epub 2008 Mar 14. PMID 18342944
- See also: Related Info — http://www.cornellneurosurgery.com
- See also: Retinoblastoma — http://mskcc.org